CLINICAL TRIAL: NCT03617705
Title: Laboratory and Field Validation of a Wrist-Worn Alcohol Monitor
Brief Title: Alcohol Monitor Validation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB201801188-N; R21AA027191 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-08-06 (Actual); Results first posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: alcohol consumption
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Alcohol Drinking | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- All participants (HIV+ and HIV- drinkers) (Other): All participants were planned to complete the BACtrack Skyn biosensor in two lab sessions, and wear the Skyn biosensor for two weeks in the field. However, due to COVID, not all participants were able to complete the lab sessions.
  Interventions: Device: Skyn Monitor Lab Session 1; Device: Skyn Monitor Field Test with EMA App; Device: Skyn Monitor Lab Session 2

INTERVENTIONS:
Device: Skyn Monitor Lab Session 1 — Participants will be instructed to wear the Skyn wrist-worn alcohol monitor and drink 3 beers over the course of an hour and a half. BrAC will be measured every 15 minutes throughout the session.
  Other Names: BACtrack Skyn; Skyn Alcohol Monitoring Device
Device: Skyn Monitor Field Test with EMA App — After Skyn Monitor Lab Session 1, participants will be instructed to wear Skyn monitor for the rest of the day and the following two weeks. Participants will also enter information on each drinking session during the two week time using a mobile-based ecological momentary assessment (EMA) to collect real-time data in daily life.
  Other Names: BACtrack Skyn; Skyn Alcohol Monitoring Device
Device: Skyn Monitor Lab Session 2 — Participants will be instructed to wear the Skyn wrist-worn alcohol monitor and drink 3 beers over the course of an hour and a half. BrAC will be measured every 15 minutes throughout the session. Participant will also complete device acceptability and usability survey.
  Other Names: BACtrack Skyn; Skyn Alcohol Monitoring Device

SUMMARY:
This study will validate a wrist-worn alcohol monitor (BACtrack Skyn) in both laboratory and real-life settings.

DETAILED DESCRIPTION:
The overarching goal of this research program is to improve alcohol intervention and eventually related clinical outcomes (e.g., liver function) among HIV+ drinkers through biosensor-assisted intervention. Research shows HIV infection can influence alcohol metabolism (i.e., higher blood alcohol levels), so it's necessary to validate the new alcohol biosensor in HIV+ drinkers rather than in general population. The primary goal of this project, as a step toward the development and evaluation of a biosensor-assisted alcohol intervention, is to validate the newly available wrist worn transdermal alcohol biosensor (BACtrack Skyn). The two specific aims are: (1) To assess validity and reliability of the Skyn biosensor using fixed-dose lab administration of alcohol through comparison with laboratory grade breathalyzer, and (2) To validate Skyn biosensor in daily life using a 2-week ecological momentary assessment (EMA) to compare self-reported drinking and the Skyn derived transdermal alcohol concentration (TAC) readings.

ELIGIBILITY:
Inclusion Criteria:

* HIV+ consumers of alcohol; self-reported ≥ 5 days with at least 1 alcoholic drink, and ≥1days with at least 3 drinks
* HIV- consumers of alcohol; self-reported ≥ 5 days with at least 1 alcoholic drink, and ≥1days with at least 3 drinks

Exclusion Criteria:

* non-drinkers
* recent addiction treatment or treatment seeking
* urine positive for illegal drugs except THC (not applicable to those who are only invited to do field test);
* past & current alcohol withdrawal
* severe alcohol use disorder (DSM-5)
* meeting criteria for current nicotine dependence (not applicable to field only participants) or current substance use disorder (excluding mild cannabis use disorder and mild/moderate alcohol use disorder)
* medical conditions (other than HIV) contraindicating alcohol
* pregnancy/breastfeeding in women
* psychosis or other severe psychiatric conditions.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yan Wang, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - HealthStreet, Gainesville, Florida
  - University of Florida, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | All Participants (HIV+ and HIV- Drinkers)
Started | 49
Completed | 40
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — lost contact after screening due to covid pandemic | 6
Not completed — withdrawal by study team due to non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants (HIV+ and HIV- Drinkers)
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (15.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 31
  Race: Black | 10
  Race: Native American | 0
  Race: Asian | 4
  Race: Multi-racial | 2
  Race: Choose not to response or no data | 2
HIV status [Count of Participants; unit: Participants]
  HIV+ | 16
  HIV- | 33

OUTCOME MEASURES:

1. Primary Outcome: Transdermal Alcohol Concentration (TAC)
Description: Here we reported mean and SD of peak TAC in the laboratory sessions and in the field test.
Time Frame: 2 weeks
Population: There were nine participants were enrolled but did not complete any study procedures due to various of reasons such as self withdrawal or administrative withdrawal, so only 40 participants had usable data for the outcome measure. Also, not all participants completed all study procedures outlined in the description due to COVID pandemic, n for lab and field data analyses varied according to how many participants completed respective study procedure.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | All Participants (HIV+ and HIV- Drinkers)
Number analyzed (Participants) | 40
ug/L
  Lab session: number analyzed (Participants) | 25
  Lab session | 38.3 (28.4)
  Field test: number analyzed (Participants) | 36
  Field test | 95.8 (113.7)

ADVERSE EVENTS:
Time Frame: Approximately 3 months
Arm/Group | All Participants (HIV+ and HIV- Drinkers)
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 0/49

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03617705/Prot_SAP_000.pdf
  • Informed Consent Form (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/05/NCT03617705/ICF_001.pdf